CLINICAL TRIAL: NCT01541254
Title: A Feasibility Study of the MicroVention,Inc.(LVIS™) Neurovascular Self-Expanding Retrievable Stent System in the Treatment of Wide-Necked Intracranial Artery Aneurysms
Brief Title: Feasibility Study of the LVIS™ (Low-profile Visualized Intraluminal Support)Device
Acronym: LVIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G110014
Record Dates: First submitted 2012-02-15; First posted 2012-02-29 (Estimated); Results first posted 2014-09-15 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Intracranial Aneurysms
Keywords: intracranial aneurysm; wide-neck; saccular; endovascular treatment; coil embolization; stent; bare platinum
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single Arm (Other): Low profile Visualized Intraluminal Device (LVIS and LVIS Jr.)
  Interventions: Device: Low profile Visualized Intraluminal Device (LVIS and LVIS Jr.)

INTERVENTIONS:
Device: Low profile Visualized Intraluminal Device (LVIS and LVIS Jr.) — Low profile Visualized Intraluminal Device (LVIS and LVIS Jr.)
  Other Names: Low-profile Vizualized Intraluminal Support Device

SUMMARY:
The purpose of this study is to evaluate the safety and probable benefit of the Low-profile Visualized Intraluminal Support (LVIS™ and LVIS™ Jr.)devices from MicroVention, Inc. when used to facilitate endovascular coiling of unruptured wide-neck intracranial aneurysms with bare platinum embolization coils.

DETAILED DESCRIPTION:
With the stent-assisted technique to treat wide neck intracranial aneurysms, the neurovascular stent is placed across the aneurysm neck, to act as a bridge to prevent coils from protruding into the parent artery. Stenting may allow to more safely achieve a higher packing density of coils. These effects may improve the rates of complete aneurysm occlusion and enhance the durability of the coiling treatment.The LVIS™ device manufactured by MicroVention, Inc. has a braided design which may provide superior conformability and parent artery apposition, as well as a more reliable continuous and uniform neck bridging than other neurovascular stents.

ELIGIBILITY:
Inclusion Criteria:

* Subject whose age is between 18 and 80 years old
* Subject with unruptured wide neck, saccular,intracranial aneurysm, < 20mm maximum diameter in any plane ( wide neck defined as neck width ≥ 4mm or dome to-neck ratio < 2).
* Subject's aneurysm arises from a parent vessel with a diameter of ≥ 2.5m and ≤ 4.5mm.
* Subject or his/her legally authorized representative understands the nature of the procedure and provides signed informed consent form.
* Subject is willing to return to the investigational site for the 30- day and 6-month follow-up evaluations

Exclusion Criteria:

* Subject who presents with ruptured aneurysm, unless rupture occured 30 days or more prior to screening.
* Subject who presents with an intracranial mass or currently undergoing radiation therapy for carcinoma of the head or neck region.
* Subject with an International Normalized Ratio (INR)≥ 1.5
* Subject with serum creatinine level >2mg/dl at time of enrollment
* Subject with known allergies to nickel-titanium metal
* Subject with known allergies to aspirin, heparin, ticlopidine, or clopidogrel
* Subject with a life threatening allergy to contrast(unless treatment for allergy is tolerated)
* Subject who has a known cardiac disorder, likely to be associated with cardioembolic symptoms such as atrial fibrillation
* Subject with any condition which in the opinion of the treating physician would place the subject at a high risk of embolic stroke
* Subject who is currently participating in another clinical research study
* Subject who has had a previous intracranial stenting procedure associated with the target aneurysm
* Subject who is unable to complete the required follow-up
* Subject who is pregnant or breastfeeding
* Subject who has participated in a drug study within the last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Fiorella, M.D., Ph.D., Principal Investigator — Stony Brook University Medical Center
Locations (6):
- United States (6):
  - Albany Medical College, Albany, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Thomas Jefferson Hospital, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern, Dallas, Texas
  - Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Fiorella D, Arthur A, Boulos A, Diaz O, Jabbour P, Pride L, Turk AS, Woo HH, Derdeyn C, Millar J, Clifton A. Final results of the US humanitarian device exemption study of the low-profile visualized intraluminal support (LVIS) device. J Neurointerv Surg. 2016 Sep;8(9):894-7. doi: 10.1136/neurintsurg-2015-011937. Epub 2015 Sep 21. PMID 26391016

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm
Started | 36
Completed | 30
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — excluded - metal allergy | 1
Not completed — enrolled after study closed | 1
Not completed — GI bleed prior to procedure | 1
Not completed — stent not required | 1
Not completed — alternate stent used | 1

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.6 (10.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Probable Benefit Measures as Successful Aneurysm Treatment With the LVIS™ Device, as Measured by Aneurysm Angiographic Occlusion of ≥ 90% at 6 Months (± 4 Weeks)
Description: Imaging from each subject to be reviewed by an independent core lab who will be comparing with baseline and post procedure images.
Time Frame: 6 months ± 4 weeks
Measure: Mean (Standard Deviation); unit: percent occlusion of aneurysm
Arm/Group | Single Arm
Number analyzed (Participants) | 28
percent occlusion of aneurysm | 95 (19)

2. Primary Outcome: Safety Measures as Any Major Stroke or Death Within 30 Days, or Major Ipsi-lateral Stroke or Neurological Death Within 6 Months
Description: A major stroke is defined as a new neurological event that persists for >24 hours and results in a ≥ 4 point increase in the National Institutes of Health Stroke Scale (NIHSS) score compared to baseline or compared to any subsequent lower score.
Time Frame: 30 days-6 months
Measure: Number; unit: patients
Arm/Group | Single Arm
Number analyzed (Participants) | 31
patients | 0 [0 to 9.2]

3. Secondary Outcome: Parent Artery Patency Measured Angiographically at 6 Months
Description: To be assessed by Independent Core Lab.
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Successful Delivery of the LVIS™ Device Measures by Technical Success
Description: Technical success being defined as: access to the lesion, successful deployment of the LVIS™ device.
Time Frame: 24 hours
Reporting Status: Not Posted

5. Secondary Outcome: Significant Stenosis(>50%) of the Treated Artery at 6 Months
Description: Parent Artery will be measured baseline and compared at 6 months post procedure per review by the Independent Core Lab.
Time Frame: 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Stent Migration at 6 Months
Description: Angiographic images will be comparing post procedure sent position to 6 months
Time Frame: 6 months
Reporting Status: Not Posted

7. Secondary Outcome: Device and Procedure Related Serious Adverse Events
Description: All Serious Adverse events will be reported per protocol
Time Frame: Day 1-6months(± 4 months)
Reporting Status: Not Posted

8. Secondary Outcome: Unplanned Embolization Coiling Within 6 Months
Description: If the target lesion(aneurysm)treated needed further embolization within 6 months of initial treatment(detected during follow up or unscheduled visit ),data will be recorded and analyzed.
Time Frame: Day 1-6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Single Arm
Serious Adverse Events (participants affected / at risk) | 1/31
Other Adverse Events (participants affected / at risk) | 8/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=31)
Stroke/TIA (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=31)
Headache (General disorders) | 8
Hematoma at access site (General disorders) | 2
Stroke or TIA (General disorders) | 2 — non-serious
Nausea (General disorders) | 2
Infection (Infections and infestations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
As part of a multi-center study the results of the national Trial shall be published by a National Principal Investigator within 12 months of completion of last study site. If no publication within that time frame, Principal Investigator is free to publish. Copies of proposed publication must be submitted to Sponsor at least 30 days in advance to ensure removal of proprietary or confidential information.